CLINICAL TRIAL: NCT01334775
Title: Comparison of Cousin Biotech® Adhesix™ Versus Conventional Mesh in Open Anterior Inguinal Hernia Repair: a Multi-centre, Randomised, Double-blinded, Controlled Clinical Trial.
Brief Title: Comparison of Self-adhering Mesh and Conventional Mesh in Inguinal Hernia Repair.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion speed too slow, no longer relevant and takeover
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Orbis Medical Centre (Other); VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL36322.068.11
Record Dates: First submitted 2011-04-05; First posted 2011-04-13 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2011-04

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia; Postoperative pain; Surgical mesh
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental - Cousin Biotech Adhesix (Experimental): Placement of a self-adhering (sutureless) surgical mesh in open anterior inguinal hernia repair
  Interventions: Procedure: Open anterior inguinal hernia repair
- Conventional - Cousin Biotech Biomesh P8 (Active Comparator): Placement of the conventional (sutured) surgical mesh in open anterior inguinal hernia repair
  Interventions: Procedure: Open anterior inguinal hernia repair

INTERVENTIONS:
Procedure: Open anterior inguinal hernia repair — Placement of a surgical mesh in open anterior inguinal hernia repair.
  Other Names: Cousin Biotech Adhesix; Cousin Biotech Biomesh P8

SUMMARY:
Inguinal hernia repair coincides with a high rate of postoperative pain, extending to over a year in 10-20% of patients. Although this is of major concern, early postoperative pain also has an important impact on patients and their ability to regain normal work and activities. Since inguinal hernia repair is the most frequently performed operation worldwide, a small reduction in loss of workdays can already have significant impact on financial issues. As for the origin of the pain, it might be the result of local inflammation caused by the mesh material, but also by nerve entrapment due to fixation techniques. The development of a new mesh which enables sutureless fixation, Cousin Biotech® Adhesix™, may overcome pain related to fixation techniques used in the open hernia repair procedure according to Lichtenstein. Furthermore, the Cousin Biotech® Adhesix™ mesh has already been in use in our institutions and surgeons familiarized themselves with the application.

The investigators would like to conduct a multicentre randomised controlled clinical trial to compare the difference in early postoperative pain after unilateral primary inguinal hernia repair in males. The procedures will be performed in day surgery. Early postoperative pain is defined as the pain during the first month, with a special interest in the first two weeks. In addition, the investigators want to measure the possible benefit in terms of time to return to work, daily activities, quality of life, operation length, complications and long term postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Primary, unilateral inguinal hernia
* Age ≥18 years
* Social status: professionally employed
* ASA-score I-III
* Signed informed consent
* Elective surgery

Exclusion Criteria:

* Female
* Bilateral and/or recurrent inguinal hernia
* Femoral or scrotal hernia
* Vasectomy
* Social status: unemployed
* Chronic use of pain medication
* Symptomatic acute hernia (i.e. bowel obstruction, incarceration, strangulation, peritonitis or perforation of bowel contents)
* ASA-score IV or above
* Incapacitated adult or no signed informed consent
* Patient is unable to speak Dutch

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Difference in early postoperative pain scores | 0-4 weeks after surgery
  Measured with VAS-scores

SECONDARY OUTCOMES:
Difference in long-term postoperative pain scores | 4 weeks - 12 months after surgery
  Measured with VAS-scores
Number of days to return to normal daily activities | 0-12 months after surgery
Number of days to return to work | 0-12 months after surgery
Differences in use of analgesics | 0-12 months after surgery
  Measured: frequency, dose and type.
Differences in reported Quality of life | 0-12 months after surgery
  Measured with SF-36 questionnaire
Number of patients with complications/adverse events | 0-12 months after surgery
  All adverse events/complications are recorded (i.e. infection, recurrence, bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole D. Bouvy, MD, PhD, Principal Investigator — Maastricht University Medical Centre, dept. of General Surgery
Locations (4):
- Netherlands (4):
  - Academic Medical Centre Amsterdam, dept. of Surgery, Amsterdam
  - Maastricht University Medical Centre, dept. of General Surgery, Maastricht
  - Orbis Medical Centre, Sittard-Geleen
  - VieCuri Medical Centre, dept. of General Surgery, Venlo